CLINICAL TRIAL: NCT05520710
Title: Symptom-Targeted Rehabilitation for Concussion in Canadian Armed Forces Veterans
Brief Title: Symptom-Targeted Rehabilitation for Concussion
Acronym: STAR-C2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Atlas Institute for Veterans and Families (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15032
Record Dates: First submitted 2022-08-19; First posted 2022-08-30 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2024-09

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Cognitive Rehabilitation; Cognitive Functioning
MeSH Terms: conditions — Brain Concussion | interventions — Cognitive Training; Educational Status

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to either the Therapy (n=30) or Education Group (n=30). At the conclusion of therapy (for the Therapy Group) or after three weeks (for the Education Group), participants will be re-administered the outcome measures. The outcome measures using the Acceptability of Intervention Measure (AIM), Intervention Appropriateness Measure (IAM), and Feasibility of Intervention Measure (FIM) will then be compared during data analysis between the two groups.
Who Masked: Outcomes Assessor
Masking Description: Assessor will be blinded to randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapy Group (Experimental): The Therapy Group will receive 6-10 individual sessions of 30-60 minutes each, delivered by a trained Occupational Therapist or Speech-Language Pathologist. The therapy will be delivered over a 4-week timeframe, with the total number of sessions per participant depending on the number of sessions needed to achieve their treatment targets. Each participant in the Therapy Group will identify three cognitive targets for treatment. Progress in reaching those targets will be documented using Goal Attainment Scaling (GAS)
  Interventions: Behavioral: Cognitive Rehabilitation
- Educational Group (Active Comparator): The education group will receive information about self-management of cognitive symptoms at the time of randomization, a common intervention for adults with mild Traumatic Brain Injury.
  Interventions: Other: Education

INTERVENTIONS:
Behavioral: Cognitive Rehabilitation — A strategy-focused intervention aimed at improving everyday cognitive function, structured to maximize treatment dose over a short time period. The shorter time period of the treatment therapy is relative to the one and only current randomized controlled trial of cognitive rehabilitation for military mTBI, the Study of Cognitive Rehabilitation Effectiveness (SCORE).
  Arms: Therapy Group
Other: Education — Educational materials, designed to help people with traumatic brain injury manage their everyday cognitive challenges will be provided through Zoom video conferencing software.
  Arms: Educational Group

SUMMARY:
The investigators are comparing two methods for helping improve everyday cognitive functioning in Canadian Armed Forces (CAF) veterans who have sustained a mild traumatic brain injury (mTBI). The two methods are 1) providing educational materials (Education Group) and 2) individual cognitive rehabilitation delivered by a trained Occupational Therapist or Speech-Language Pathologist (Therapy Group). The study is a pilot randomized controlled clinical trial (RCT), and will serve as pilot data for a future RCT.

DETAILED DESCRIPTION:
The investigators are comparing two different methods for helping Canadian Armed Forces veterans with mild traumatic brain injury (mTBI) manage everyday cognitive difficulties. Cognitive rehabilitation is a type of therapy that helps people with brain injury who have challenges in everyday thinking. The investigators have developed a streamlined version of this type of cognitive rehabilitation therapy that can be done in person or virtually and takes place over a 3-week period. The investigators will provide education materials only to one group and individual cognitive rehabilitation delivered by a trained Speech Language Pathologist or Occupational Therapist to the other group. The investigators want to find out whether the individual therapy is better than providing the usual educational material. The therapy sessions are audio-recorded. At McMaster, the investigators job is to listen to the recordings and making sure the therapists are following the study manual. That includes making notes of what the therapists say or do. What the investigators learn in this study may help veterans with mTBI and cognitive issues affect their abilities to do everyday activities.

ELIGIBILITY:
Inclusion Criteria:

* Is a community-dwelling Canadian Armed Forces veteran.
* Is age 18 years or older.
* Self-identifies as a fluent English speaker.
* Has no previous history of neurological disorder affecting cognition, by self-report.
* Is able to participate in rehabilitation for 4 weeks: 3 weeks of treatment + baseline + outcome assessment, with potential rescheduling for missed sessions.
* Is not actively participating in cognitive rehabilitation directed by a registered health professional (e.g., speech-language pathologist or occupational therapist).
* Has access to an electronic device with Zoom video platform capacity and internet access.

Exclusion Criteria:

* A score of less than 20 on the Montreal Cognitive Assessment (MoCA), which indicates a risk for dementia.
* Cannot identify at least 3 problems on the Common Cognitive Complaints after Concussion Questionnaire (C4), as there would be insufficient areas for intervention.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Recruitment Rate | 12 months
  The primary outcome is the rate of recruitment, average 5 per month. The primary outcome is the rate of recruitment and retention rate reported as total number of participants recruited and retained.
Adherence to Intervention | 12 months
  Three quarters of participants should complete 80% of the prescribed intervention

SECONDARY OUTCOMES:
Acceptability of the Intervention | Measures administered during intake (baseline), immediately after one of sessions 6-10 depending on targets achieved, and 1 month post-treatment.
  The acceptability will be assessed by clinicians and participants. At least three quarters of participants and clinicians will provide a rating of 4 on the Acceptability of Intervention Measure (AIM).
Acceptability of the Appropriateness | Measures administered during intake (baseline), immediately after one of sessions 6-10 depending on targets achieved, and 1 month post-treatment.
  The acceptability will be assessed by clinicians and participants. At least three quarters of participants and clinicians will provide a rating of 4 on the Intervention Appropriateness Measure (IAM).
Acceptability of the Feasibility | Measures administered during intake (baseline), immediately after one of sessions 6-10 depending on targets achieved, and 1 month post-treatment.
  The acceptability will be assessed by clinicians and participants. At least three quarters of participants and clinicians will provide a rating of 4 on the Feasibility of Intervention Measure (FIM).

CONTACTS AND LOCATIONS:
Overall Officials: Lyn Turkstra, PhD, Principal Investigator — McMaster University School of Rehabilitation Science; Jackie Bosch, PhD, Principal Investigator — McMaster University School of Rehabilitation Science
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garber BG, Rusu C, Zamorski MA. Deployment-related mild traumatic brain injury, mental health problems, and post-concussive symptoms in Canadian Armed Forces personnel. BMC Psychiatry. 2014 Nov 20;14:325. doi: 10.1186/s12888-014-0325-5. PMID 25410348
- [Background] Soble JR, Silva MA, Vanderploeg RD, Curtiss G, Belanger HG, Donnell AJ, Scott SG. Normative Data for the Neurobehavioral Symptom Inventory (NSI) and post-concussion symptom profiles among TBI, PTSD, and nonclinical samples. Clin Neuropsychol. 2014;28(4):614-32. doi: 10.1080/13854046.2014.894576. Epub 2014 Mar 14. PMID 24625213
- [Background] Tanev KS, Pentel KZ, Kredlow MA, Charney ME. PTSD and TBI co-morbidity: scope, clinical presentation and treatment options. Brain Inj. 2014;28(3):261-70. doi: 10.3109/02699052.2013.873821. PMID 24568300
- [Background] Hoffman AN, Taylor AN. Stress reactivity after traumatic brain injury: implications for comorbid post-traumatic stress disorder. Behav Pharmacol. 2019 Apr;30(2 and 3-Spec Issue):115-121. doi: 10.1097/FBP.0000000000000461. PMID 30640181
- [Background] Management of Concussion/mTBI Working Group. VA/DoD Clinical Practice Guideline for Management of Concussion/Mild Traumatic Brain Injury. J Rehabil Res Dev. 2009;46(6):CP1-68. No abstract available. PMID 20108447
- [Background] Loignon A, Ouellet MC, Belleville G. A Systematic Review and Meta-analysis on PTSD Following TBI Among Military/Veteran and Civilian Populations. J Head Trauma Rehabil. 2020 Jan/Feb;35(1):E21-E35. doi: 10.1097/HTR.0000000000000514. PMID 31479073
- [Background] Cicerone KD, Goldin Y, Ganci K, Rosenbaum A, Wethe JV, Langenbahn DM, Malec JF, Bergquist TF, Kingsley K, Nagele D, Trexler L, Fraas M, Bogdanova Y, Harley JP. Evidence-Based Cognitive Rehabilitation: Systematic Review of the Literature From 2009 Through 2014. Arch Phys Med Rehabil. 2019 Aug;100(8):1515-1533. doi: 10.1016/j.apmr.2019.02.011. Epub 2019 Mar 26. PMID 30926291
- [Background] Marshall S, Bayley M, McCullagh S, Velikonja D, Berrigan L, Ouchterlony D, Weegar K; mTBI Expert Consensus Group. Updated clinical practice guidelines for concussion/mild traumatic brain injury and persistent symptoms. Brain Inj. 2015;29(6):688-700. doi: 10.3109/02699052.2015.1004755. Epub 2015 Apr 14. PMID 25871303
- [Background] Cooper DB, Bowles AO, Kennedy JE, Curtiss G, French LM, Tate DF, Vanderploeg RD. Cognitive Rehabilitation for Military Service Members With Mild Traumatic Brain Injury: A Randomized Clinical Trial. J Head Trauma Rehabil. 2017 May/Jun;32(3):E1-E15. doi: 10.1097/HTR.0000000000000254. PMID 27603763
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Malec JF, Smigielski JS, DePompolo RW. Goal attainment scaling and outcome measurement in postacute brain injury rehabilitation. Arch Phys Med Rehabil. 1991 Feb;72(2):138-43. PMID 1991015
- [Background] Blevins CA, Weathers FW, Davis MT, Witte TK, Domino JL. The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress. 2015 Dec;28(6):489-98. doi: 10.1002/jts.22059. Epub 2015 Nov 25. PMID 26606250
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- See also: The Canadian Occupational Performance Measure — https://www.thecopm.ca/